CLINICAL TRIAL: NCT01689168
Title: Chiropractic Treatment With Counseling Versus Counseling Alone for Promoting Smoking Cessation: A Randomized Clinical Trial
Brief Title: Chiropractic Treatment With Counseling Versus Counseling Alone for Promoting Smoking Cessation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ran out
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, KevinRose, Professor, Southern California University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROSE004
Record Dates: First submitted 2012-06-05; First posted 2012-09-21 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Counseling; Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling plus chiropractic adjustments (Experimental)
  Interventions: Behavioral: Counseling; Procedure: Chiropractic adjustment
- Counseling alone (Active Comparator)
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Tobacco cessation counseling
Procedure: Chiropractic adjustment — Full spine high velocity, low amplitude manipulation of the spine
  Arms: Counseling plus chiropractic adjustments

SUMMARY:
Tobacco use is the number one killer of Americans today. Most current smokers have tried and failed to quit at least once. Smokers are addicted to the nicotine in tobacco products, and withdrawal from smoking can lead to physical symptoms such as irritability, anxiety, nervousness, depression and insomnia.

This study will examine the effects of tobacco cessation counseling and chiropractic treatments on smokers who desire to quit.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 yrs and above
* Smokers with desire to quit smoking

Exclusion Criteria:

* Received chiropractic treatment or other manipulative therapies within the last month
* Have received any therapy for smoking cessation during the last month
* Visceral, systemic or joint inflammatory disease
* A history of low back surgery
* Osteoporosis
* Prolonged systemic corticosteroid medication
* Pregnancy
* Recent spinal fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Tobacco cessation | Smoking diary will be complete for 3 months
  Has the subject quit smoking?
Urinary cotinine | Baseline, 14, 30, 60 and 90 days
  An urinary test for nicotine metabolites

SECONDARY OUTCOMES:
Blood pressure | Baseline, 14, 30, 60 days
Weight | Baseline, 14, 30, 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Rose, DC, MPH, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- University Health Center - Whittier, Whittier, California, United States